CLINICAL TRIAL: NCT00208260
Title: Randomized Phase II Trial Followed by Phase III Trial With Molecular Biology Study, Comparing a Standard Bi-therapy vs 3 Arms of Intensified Chemotherapy in Patients With Unresectable or Not Optimally Resectable Colorectal Cancer Liver Metastases.
Brief Title: Intensified Chemotherapy in CRC After Resection of Liver Metastases
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Collaborators: Pfizer (Industry); Sanofi (Industry); Chugai Pharmaceutical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METHEP/2004/22
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Cancer; Liver Metastases; Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — IFL protocol; Folfox protocol; folfirinox

ARMS (5):
- A (Active Comparator): FOLFIRI
  Interventions: Drug: FOLFIRI
- B (Active Comparator): FOLFOX-4
  Interventions: Drug: FOLFOX-4
- C (Experimental): FOLFIRI-HD
  Interventions: Drug: FOLFIRI-HD
- D (Experimental): FOLFOX-7
  Interventions: Drug: FOLFOX-7
- E (Experimental): FOLFIRINOX
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRI — FOLFIRI : Irinotecan : 180 mg/m² 90 min continuous perfusion during levorin d1 every 2 weeks
  Arms: A
Drug: FOLFOX-4 — FOLFOX 4 : Oxaliplatine : 85 mg/m² 2h continuous perfusion during levorin d1 every 2weeks
  Arms: B
Drug: FOLFIRI-HD — High Dose FOLFIRI : Irinotecan : 260 mg/m² in 90min continuous perfusion during levorin d1 every 2 weeks
  Arms: C
Drug: FOLFOX-7 — FOLFOX 7 : Oxaliplatine : 130 mg/m² in 2h continuous perfusion during levorin d1 every 2 weeks
  Arms: D
Drug: FOLFIRINOX — FOLFIRINOX : Oxaliplatine : 85 mg/m² 2h continuous perfusion followed by 1H rest followed by 90 min continuous perfusion of irinotecan : 180 mg/m² during levorin d1 every 2 weeks
  Arms: E

SUMMARY:
Randomized, open label, multicentre phase II trial followed by phase III comparing overall survival after having selected the best experimental arm.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven adenocarcinoma of the colon or rectum without previous resection, or clinically asymptomatic (with or without stent)
* Hepatic unresectable metastases R0: due to close vascular contact, or due to liver remaining mass less than 25 to 30 % of functional liver.
* Not optimally resectable metastases
* Extra-hepatic disease will be accepted in case of: asymptomatic primary tumour or tumor requiring no urgent surgery (in less than 3 months); three of less than three lung metastases (thoracic scan diameter less than 2 cm) and potentially respectable.
* Synchronous and metachronous hepatic metastases
* WHO performance status 0-1
* Adjuvant chemotherapy allowed, except oxaliplatin and irinotecan based combination.
* No prior treatment of the liver metastases, whatever.
* Life expectancy equal or more than 3 months

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2004-04; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Response | end of chemotherapy

SECONDARY OUTCOMES:
Safety | during study treatment
Survival | 2 years
Secondary resection | surgery after chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Marc YCHOU, MD, PhD, Principal Investigator — CRLC Val d'Aurelle; Michel RIVOIRE, MD, Study Chair — CRLC Leon Berard - Lyon
Locations (1):
- CRLC Val d'Aurelle, Montpellier, France

REFERENCES:
- [Result] Ychou M, Rivoire M, Thezenas S, Quenet F, Delpero JR, Rebischung C, Letoublon C, Guimbaud R, Francois E, Ducreux M, Desseigne F, Fabre JM, Assenat E. A randomized phase II trial of three intensified chemotherapy regimens in first-line treatment of colorectal cancer patients with initially unresectable or not optimally resectable liver metastases. The METHEP trial. Ann Surg Oncol. 2013 Dec;20(13):4289-97. doi: 10.1245/s10434-013-3217-x. Epub 2013 Aug 17. PMID 23955585